CLINICAL TRIAL: NCT04847323
Title: Clinical Effectiveness of Bonded Versus Vacuum-formed Retainers After 12 Months: A Randomized Controlled Trial
Brief Title: Clinical Effectiveness of Bonded Versus Vacuum-formed Retainers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Silvio Augusto Bellini-Pereira, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22092919.7.0000.5417; 001 (Other Grant/Funding Number: Coordination for the Improvement of Higher Educational Personnel)
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Relapse
Keywords: Orthodontic Retainers; Orthodontic Appliances, Removable; Orthodontics
MeSH Terms: conditions — Recurrence | interventions — Orthodontic Appliances, Fixed

STUDY DESIGN:
Intervention Model Description: This was a 2-arm parallel randomized controlled trial. Therefore, the selected patients were randomly divided into two groups.
  Group 1: Bonded V-bend retainers. Group 2: Vacuum-formed retainers. Randomization was performed through sequentially numbered, opaque envelopes prepared by a colleague independent of the study.
Who Masked: Outcomes Assessor
Masking Description: Masking of the principal investigator and participants was not be possible due to the nature of the interventions. Nonetheless, the outcome assessor was blinded for the periodontal and patient perception variables.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- V-bend Bonded Retainer (Active Comparator): The V-bend retainer was bonded in the lingual surface of the anterior teeth. The retainer was constructed using 0.024" stainless steel wires. Differently from the conventional bonded retainers, this retainer presents V-bends in the sagittal direction, parallel to the occlusal plane in each interproximal contact point of the incisors and canines.
  The retainers was bonded after adequate etching with phosphoric acid and application of adhesive with a low viscosity resin.
  Interventions: Device: V-bend Bonded Retainer
- Vacuum-formed Retainer (Active Comparator): The removable Vacuum-formed retainers were made of acetate 1mm thickness. They were made at the same appointment of debonding using plaster models. The patients were instructed to use the retainers only during nights.
  Interventions: Device: Vacuum-formed Retainer

INTERVENTIONS:
Device: V-bend Bonded Retainer — Traditional stainless steel retainer commonly bonded in the anterior teeth of the mandibular arch to maintain their alignment after orthodontic treatment.
  Other Names: Bonded Retainer; Canine-to-Canine Retainer; Fixed Retainer
  Arms: V-bend Bonded Retainer
Device: Vacuum-formed Retainer — Removable retainers made of plastic and derivatives. Currently gaining popularity due to the increased use of esthetic aligners. These clear retainers have the objective to maintain stable the results obtained after orthodontic treatment. They cover all the surfaces of the teeth up to the first or second molars.
  Other Names: Thermoplastic Retainer; Clear Retainer
  Arms: Vacuum-formed Retainer

SUMMARY:
The purpose of the study was to compare the clinical effectiveness of bonded versus vacuum-formed retainers regarding their retention capacity; periodontal health; survival rates; and patients' perception after 12 months of removal of fixed appliances.

The null hypotheses considered that there was no differences between the retainers in relation to the aspects evaluated.

DETAILED DESCRIPTION:
This single-center randomized controlled trial was performed at the Department of Orthodontics, Bauru Dental School, University of São Paulo, Brazil.

A total of 50 patients completing orthodontic treatment were recruited. The patients were prospectively and randomly allocated into two groups. The first group consisted of 25 patients with canine-to-canine V-bend bonded retainers; while the second group comprised 25 patients with vacuum-formed retainers. In both groups, the same retainers were installed in the maxillary and mandibular arches.

Patients were evaluated at deboning (T0), after 3 months (T1), 6 months (T2), and 12 months (T3). In each appointment, digital models were obtained and the other clinical variables were evaluated. The primary and secondary outcomes were compared between retainers in the time-points evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the proper completion of orthodontic treatment and correction of the initial malocclusion.
* Acceptable oral hygiene (assessed through clinical examination).
* Presence of all teeth up to the second molars.
* Clinically acceptable teeth alignment.

Exclusion Criteria:

* Patients with any systemic condition that may have an influence on periodontal health.
* Patients with facial deformities.
* Initial malocclusion that required extreme corrections, large transverse expansions or orthognathic surgery.
* History of periodontal diseases.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Changes in Little Irregularity Index (LII) | Changes were compared at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Stability was evaluated comparing the changes in the Little Irregularity Index (LII) between time-points. The average of the linear distances between the anatomical contact points of the anterior teeth were considered.

SECONDARY OUTCOMES:
Intercanine Distance | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Distance between the cusp tips of the right and left permanent canines. In the maxilla and mandible.
Intermolar Distance | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Distance between the tips of the mesiobuccal cusps of the first right and left permanent molars. In the maxilla and mandible.
Overjet | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Distance between the incisal edge of the maxillary central incisor and the incisal edge of the mandibular incisor, parallel to the occlusal plane.
Overbite | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Distance between the incisal edge of the upper central incisor and the incisal edge of the lower incisor, perpendicular to the occlusal plane.
Calculus Accumulation | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Periodontal status was evaluated regarding the amount of calculus accumulation using the Simplified Oral Hygiene Index from Greene and Vermillion, 1978. The extension of calculus was estimated visually in all erupted teeth. Each teeth received a score ranging from 0 to 3. Minor scores indicated absence of calculus while higher scores indicated greater calculus accumulation on the tooth surfaces.
Gingival Health | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Periodontal status was evaluated regarding the patients' gingival health using the Gingival Index described by Loe, 1967. The gingival health was estimated clinically with a periodontal probe in all erupted teeth. Each teeth received a score ranging from 0 to 3. Minor scores indicated acceptable gingival health while higher scores indicated greater inflammation and unacceptable gingival health.
Plaque Accumulation | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Periodontal status was evaluated regarding the amount of plaque accumulation using the Plaque Index from Loe, 1967. The extension of plaque was estimated clinically using a periodontal probe in all erupted teeth. Each teeth received a score ranging from 0 to 3. Minor scores indicated absence of plaque while higher scores indicated greater plaque accumulation on the tooth surfaces.
Retainers Survival Rates | Evaluation was performed during the 12 Months of follow-up.
  The number and cause of failures for each patient was recorded during the 12-month follow-up. From these data, the total survival rate of the retainers was estimated as a percentage, as well as its major causes of failure.
Patients' Perception | Evaluation was performed at T0 (Debonding); T1 (3 Months Follow-up); T2 (6 Months Follow-up); and T3 (12 Months Follow-up).
  Patients' perception was assessed using a Visual Analogue Scale (VAS) containing a questionnaire with 9 questions related to the use of the retainers. Each question received a score ranging from 0 to 10. Minor scores indicated that the patient felt extremely uncomfortable during the retention period while higher scores indicated that the patients felt highly comfortable.

CONTACTS AND LOCATIONS:
Locations (1):
- Bauru Dental School, University of São Paulo, Bauru, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No